CLINICAL TRIAL: NCT01764672
Title: Effects of Methylphenidate on Resting State Connectivity in Healthy Controls and in Adults With Attention Deficit Hyperactivity Disorder.
Brief Title: Effect of Methylphenidate on Connectivity
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Iris Sommer (Other)
Collaborators: Netherlands Brain Foundation (Other)
Responsible Party: Sponsor-Investigator, Iris Sommer, Prof.Dr., UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-005339-95; NL42603.041.12 (Registry Identifier: Toetsingonline)
Record Dates: First submitted 2012-12-21; First posted 2013-01-09 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Healthy Adults; Methylphenidate; Functional connectivity; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Deficit Hyperactivity Disorder (Experimental): Adult males with Attention Deficit Hyperactivity disorder will participate in a crossover design and receive both methylphenidate and placebo on two separate days.
  Interventions: Drug: Methylphenidate; Other: Placebo
- Healthy adults (Experimental): Healthy male adults will participate in a crossover design and receive both methylphenidate and placebo on two separate days.
  Interventions: Drug: Methylphenidate; Other: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Oral dose 40mg (2 x 20mg)
  Other Names: Ritalin
Other: Placebo — Oral intake of 2 placebo tablets

SUMMARY:
The goal of the study is to use graph theory to examine how the organization of the functional brain network may be altered by the administration of methylphenidate. This effect is to be compared between methylphenidate intake and placebo intake, as well as between healthy adult males and adult males with a diagnosis of Attention Deficit Hyperactivity Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Written informed consent
* For the Attention Deficit Hyperactivity Disorder group only: a diagnosis of Attention Deficit Hyperactivity Disorder

Exclusion Criteria:

* Age under 18 or > 40
* Previous or current medical, psychiatric, or neurological problems (with exception of Attention Deficit Hyperactivity Disorder group)
* Use of psychotropic medication
* Use of recreational drugs in the two weeks before start of the study
* Consuming an equivalent of > 5 cups of coffee per day
* Consuming three or more alcohol units per day
* The presence of one or more of the contraindications or warnings against the study drug as listed in the Summary of Product Characteristic
* Presence of any contraindication to Magnetic Resonance Imaging scanning (e.g. implanted metallic object or electronic device)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
The difference in functional connectivity as measured with functional Magnetic Resonance Imaging between participants who ingested methylphenidate and those who ingested placebo. | After the last patient has completed the last visit, which is expected to be two years after the start of the study
  The primary objective in the current trial is to use graph theory to examine how the organization of the functional brain network may be altered by the administration of methylphenidate. The main question we intend to answer in this study, is whether, and if so to what extent, methylphenidate affects the organization of brain networks.

SECONDARY OUTCOMES:
The difference in functional connectivity as measured by functional Magnetic Resonance Imaging between participants with Attention Deficit Hyperactivity Disorder and healthy controls. | After the last patient has completed the last visit, which is expected to be two years after the start of the study
  To examine if any of the effects on brain connectivity differ between participants with Attention Deficit Hyperactivity Disorder versus healthy controls.
The correlation of graph metrics (as a measure of functional network organization) with performance (scores) on cognitive tasks and blood levels of methylphenidate. | After the last patient has completed the last visit, which is expected to be two years after the start of the study
  To examine how a reorganization of brain networks as described in the primary objective is related to improvements in cognitive performance and to blood levels of methylphenidate.
The correlation of whole brain cortical thickness and white matter volume as measured with Magnetic Resonance Imaging with both graph metrics as measured with functional Magnetic Resonance Imaging and scores on cognitive tests. | After the last patient has completed the last visit, which is expected to be two years after the start of the study
  To examine if certain network structures of the brain, such as cortical thickness and white matter volume, are related to susceptibility to medication efficacy and if the structural qualities are related to cognitive performance.

CONTACTS AND LOCATIONS:
Overall Officials: Iris EC Sommer, Prof, Dr., Study Director — UMC Utrecht; Martijn P Van den Heuvel, Dr., Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands